CLINICAL TRIAL: NCT04784819
Title: Cross-cultural Adaptation, Reliability and Validity of the Occupational Balance-Questionnaire (OB-Quest) in Turkish
Brief Title: Turkish Version of Occupational Balance-Questionnaire (OB-Quest)
Acronym: OB-QUEST
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Collaborators: Hacettepe University (Other); Istanbul Kültür University (Other); Ondokuz Mayıs University (Other); Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ZEYNEP BAHADIR AGCE, Assistant Professor, Uskudar University
Other Study IDs: GO 15/735-43
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Occupational Balance; Occupational Therapy; Survey; Assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study was to translate and culturally adapt the Occupational Balance Questionnaire (OB-Quest) and evaluate the psychometric properties of the translated version by validity and reliability testing.

DETAILED DESCRIPTION:
This study consists of two parts; in the first part, the translation and cross-cultural adaptation were undertaken, and in the second part, analyses of psychometric properties of OB-Quest Turkish were performed.

Part I: Translation and cross-cultural adaptation

The developers of the original questionnaire were contacted to seek their permission to translate the OB-Quest into Turkish and permission was obtained by the researchers via email. The five-stage translation-back translation method proposed by Beaton et al were used in the cross-cultural adaptation of the questionnaire (Beaton et al., 2000).

The first stage included translation procedures, and two therapists translated the questionnaires' English form into Turkish. In the second stage, two translations were compared to avoid any discrepancy and converted a single text by the research team. Generally, OB-Quest has a simple and understandable sentence structure. Therefore, it did not require any cultural adaptation, simple arrangement was enough to provide clarity. Researchers arranged on the last two items. These items consisting of a single sentence were divided into two as 'example and question', to overcome the complexity of the questions and maintain the integrity of the meaning. After the corrections, researchers had an agreement on the Turkish version of OB-Quest. In the third stage, the back translation of the final text from Turkish to English was made by two native English speakers whose Turkish very well. In the fourth step, the researchers compared the original text with the last English form and produced the final version. The final stage covered the pilot study to get understanding items. After the translation process was completed, a pilot study was conducted with a group of 30 people. Participants approved the final version was appropriate and understandable. The participants in the pilot study did not include in the sample group.

Part II Analysis of the psychometric properties of OB-Quest

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years
* native speakers of Turkish
* literate of Turkish
* healthy
* volunteered to participate in the study

Exclusion Criteria:

* diagnosed with acute/chronic disease

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study conducted with people who were in the Department of Health Science at the University and their relatives between April 2018 to May 2020. Students, patients, faculty staff or their relatives were invited to the study, those who met the inclusion criteria, and volunteers were asked to complete the forms.
Sampling Method: Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Occupational Balance-Questionnaire (OB-Quest) | 5 minutess.
  OB-Quest was developed by Dür et all., as a self-reported outcome instrument to evaluate occupational balance. It was developed based on the experiences of chronic patients and healthy people. The OB-Quest original version internal consistency was shown by Cronbach's alpha as 0.57. It has consisted of ten items and seven components: challenging and relaxing activities; accepted activities; impact of health status on activities; stress, rest and sleep; various activities; and adaptation of activities according to changing living conditions. Each item is scored on a Likert scale ranging from 1 to 3, where 1 indicates a positive score such as 'having a wide variety of activities, and 3 indicates a negative score such as 'not having a wide variety of activities or not showing any variation'. A low score is interpreted as a good occupational balance (Dür et al., 2014).

SECONDARY OUTCOMES:
The Beck Depression Inventory (BDI) | 15 minutes
  Beck Depression Inventory was developed by Beck in 1961. It includes 21 items that measure the level of depressive symptoms. Each item contains a four-grade self-assessment that determines depression-specific behavior (Beck, 1961). High scores represent an increase in depressed states. The Turkish scale was adapted by Hisli et al. (Hisli Şahin, 1988).
The 12-item Short Form Survey (SF-12) | 7 minutes
  SF-12 was created by simplifying SF-36. It was developed by Ware et al. in 1993 to evaluate quality of life and health outcomes (Ware Jr et al., 1996). SF-12 scores were calculated for each SF-12 physical (SF-12 PCS) and SF-12 mental (SF-12 MCS) component and added to determine the overall score according to the algorithm described by Ware et al. low scores are associated with low quality of life (Ware et al., 1995). It is an easy-to-apply questionnaire with proven reliability and validity in Turkish (Kocyigit et al., 1999).

CONTACTS AND LOCATIONS:
Overall Officials: ZEYNEP BAHADIR AGCE, PHD, Study Director — occupational therapy
Locations (1):
- Zeynep Bahadir Agce, Istanbul, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dur M, Steiner G, Fialka-Moser V, Kautzky-Willer A, Dejaco C, Prodinger B, Stoffer MA, Binder A, Smolen J, Stamm TA. Development of a new occupational balance-questionnaire: incorporating the perspectives of patients and healthy people in the design of a self-reported occupational balance outcome instrument. Health Qual Life Outcomes. 2014 Apr 5;12:45. doi: 10.1186/1477-7525-12-45. PMID 24708642